CLINICAL TRIAL: NCT03147690
Title: A Multicenter Trial of Contrast-Enhanced Ultrasound in the Evaluation of Abdominal Solid Organ Injuries in Pediatric Trauma
Brief Title: Contrast-Enhanced Ultrasound in the Evaluation of Abdominal Injuries in Children
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped for futility
Sponsor: David Mooney (Other)
Responsible Party: Sponsor-Investigator, David Mooney, Director Trauma Program, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P00025242
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Injury
Keywords: Solid Organ Injury
MeSH Terms: conditions — Abdominal Injuries | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Study Participants (Experimental): All subjects will have an abdominal non-contrast ultrasound performed. Lumason will then be administered at a dose of 0.03mL/kg up to a maximum dose of 2.4mL and a contrast-enhanced ultrasound will be performed. The dose will be given twice, for a total maximum dose per subject of 4.8mL
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — Lumason will be administered at a dose of 0.03 mL/kg up to a maximum dose of 2.4mL injected into a peripheral intravenous catheter. An abdominal contrast enhanced ultrasound will be performed to look for solid organ injury. The will be given twice during the intervention, for a total maximum dose per subject of 4.8mL.
  Other Names: SonoVue

SUMMARY:
This study proposes to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) in diagnosing abdominal solid organ injuries in pediatric patients. 146 subjects will be enrolled across approximately 8 sites in the US. All subjects will have had a Computerized Tomography (CT) scan as part of standard of care, confirming at least one solid organ abdominal injury. All subjects will have an abdominal ultrasound without contrast, followed by a contrast-enhanced ultrasound using the contrast agent Lumason. Ultrasound and contrast-enhanced ultrasound results will be compared to the CT scan results. The study procedures will take place within 48 hours of injury.

DETAILED DESCRIPTION:
This is an interventional study proposes to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) in diagnosing abdominal solid organ injuries in pediatric patients. 146 subjects will be enrolled across approximately 8 sites in the US. All subjects will have had a Computerized Tomography (CT) scan as part of standard of care, confirming at least one solid organ abdominal injury. All subjects will have an abdominal ultrasound without contrast, followed by a contrast-enhanced ultrasound using the contrast agent Lumason. Ultrasound and contrast-enhanced ultrasound results will be compared to the CT scan results. The study procedures will take place within 48 hours of injury. At conclusion of enrollment of all subjects a centralized review of CT vs. CEUS will occur to compare to real time readings.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable, as determined by the trauma team
* Age 8 through 17 years
* Interpretable CT of the abdomen and pelvis that demonstrates at least one abdominal solid organ injury among the liver, spleen, pancreas, and kidneys
* Plan for observation or admission to the hospital
* Candidate for abdominal ultrasound based on body habitus
* Have a Glasgow Coma Score of 15
* Able to complete the study procedures within 48 hours of injury

Exclusion Criteria:

* Known cardiac abnormality
* Pulmonary hypertension
* Known sensitivity to sulfur hexafluoride, polyethylene glycol 4000, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), or palmitic acid
* Unable to roll over
* Unable to assent
* Pregnant
* Lactating
* CT images not available for transmission to central image repository

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mooney, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (8):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Riley Children's Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Study Participants
Started | 74
Completed | 71
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 13.3 [8.0 to 17.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 64
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients for Whom All Organs Identified by CT With Injuries Are Also Identified by CEUS, Regardless of Injury Grade.
Description: During analysis, results of contrast enhanced ultrasound will be compared to results of CT scan that was performed as part of clinical care to determine if the organs identified as injured by CT were also identified as injured by CEUS.
Time Frame: At the time the CEUS is performed, within 48 hours of injury.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 74
Participants | 53

2. Secondary Outcome: For Each Organ, the Proportion of Patients for Whom the Organ is Identified by CT and CEUS as Injured (Regardless of Grade).
Description: Results will be categorized by organ and analyzed to determine the percentage of injuries for each organ that were identified by CT that were also identified by CEUS.
Time Frame: At the time the CEUS is performed, within 48 hours of injury.
Measure: Count of Participants; unit: Participants
Groups:
- Liver: All subjects will have a liver injury identified by CT
- Spleen: All subjects will have a spleen injury identified by CT
- Right Kidney: All subjects will have a right kidney injury identified by CT
- Left Kidney: All subjects will have a left kidney injury identified by CT
- Pancreas: All subjects will have a pancreas injury identified by CT
Arm/Group | Liver | Spleen | Right Kidney | Left Kidney | Pancreas
Number analyzed (Participants) | 23 | 40 | 9 | 12 | 1
Participants | 16 | 36 | 6 | 9 | 0

3. Secondary Outcome: Proportion of Injuries Identified by CEUS Which Are Within 1 Grade of the Injury Identified by CT.
Description: The grade for the severity of the injury as determined by CEUS will be compared to the grade for the severity of the injury as determined by CT scan.
Time Frame: At the time the CEUS is performed, within 48 hours of injury.
Measure: Count of Participants; unit: Participants
Arm/Group | Liver | Spleen | Right Kidney | Left Kidney | Pancreas
Number analyzed (Participants) | 23 | 40 | 9 | 12 | 1
Participants | 11 | 34 | 4 | 9 | 0

4. Secondary Outcome: Proportion of Patients Where the Absence or Presence of Peritoneal Fluid Identified by CT is Also Identified by CEUS.
Description: The presence or absence of peritoneal fluid as determined by CEUS will be compared to the presence or absence of peritoneal fluid as determined by CT scan.
Time Frame: At the time the CEUS is performed, within 48 hours of injury.
Measure: Count of Participants; unit: Participants
Groups:
- CT-Fluid: All subjects will have fluid identified by CT
- CT-No Fluid: All subjects will have no fluid identified by CT
Arm/Group | CT-Fluid | CT-No Fluid
Number analyzed (Participants) | 55 | 19
Participants | 42 | 9

5. Secondary Outcome: Proportion of Patients With Agreement Between 'Real-time' and Centralized Interpretation of CEUS Images.
Description: The contrast-enhanced ultrasounds will be re-read by a centralized reviewer and the results compared to those from the real-time reading.
Time Frame: At the time the CEUS is performed, within 48 hours of injury.
Measure: Number; unit: percentage of participants
Groups:
- Liver; Spleen; Right Kidney; Left Kidney; Pancreas; All Organs: All subjects whose central review is complete
Arm/Group | Liver | Spleen | Right Kidney | Left Kidney | Pancreas | All Organs
Number analyzed (Participants) | 68 | 68 | 68 | 68 | 68 | 68
percentage of participants | 77.9 | 72.1 | 88.2 | 95.6 | 98.5 | 44.1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of consent until 30 minutes after the second Lumason injection, within 48 hours of the participant's injury.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 3/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=74)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03147690/Prot_SAP_002.pdf